CLINICAL TRIAL: NCT05421104
Title: Ruxolitinib for the Treatment of Polycythemia Vera in Patients Who Are Resistant to or Intolerant of Hydroxyurea: a Retrospective Non-interventional Study Using the US Optum Electronic Health Record Data Source.
Brief Title: Ruxolitinib for Polycythemia Vera in Patients Resistant to or Intolerant of Hydroxyurea.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424B3001
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Polycythemia Vera (PV)
Keywords: Polycythemia vera,; Ruxolitinib,; JAK protein inhibitor,; Hydroxyurea,; Thrombotic events
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Ruxolitinib (RUX): PV patients who were resistant to or intolerant of HU (as defined on the index date) and switched to RUX in the post-index period.
  Interventions: Other: Ruxolitinib
- Best available therapy (BAT): PV patients who were resistant to or intolerant of Hydroxyurea (HU) (as defined on the index date) and continued HU treatment or switched to other available therapies other than RUX in the post-index period.

INTERVENTIONS:
Other: Ruxolitinib — PV patients who were resistant to or intolerant of HU (as defined on the index date) and switched to RUX in the post-index period.
  Other Names: Jakavi
  Groups: Ruxolitinib (RUX)

SUMMARY:
This was an analytical and descriptive, non-interventional, retrospective cohort study of PV patients aged ≥ 18 years in the US using a secondary data source, Optum EHR database.

DETAILED DESCRIPTION:
The Optum EHR database was current up to 30-Jun-2020.

Identification period: From 01-Apr-2007 to 30-Jun-2019

Study period: From 01-Jan-2007 to 30-Jun-2020

Index date:

First evidence of resistance to or intolerance of HU treatment in patients with PV according to modified European Leukemia Net (ELN) criteria and defined as:

1. HCT ≥ 45% with phlebotomy (last phlebotomy within last 3 months) Or
2. Platelet count > 400 x 109/L and presence of palpable splenomegaly (palpable spleen up to 3 months after platelet count)

Pre-index period:

Patients had a minimum of 3 months pre-index data available. Pre-index data availability was determined using the reported 'first month active' field.

Post-index period:

There was no minimum post-index period required. Each patient had a 'first month active' and 'last month active' reported within the database. As the 'last month active' was based on any activity in the database, including encounters such as letters and emails which occurred several months after the 'death_date' of the patient, using the 'last month active' can overestimate the follow-up for a given patient. For this reason, the end of follow-up for each patient was defined as the date of the last activity within the diagnosis, observations, prescriptions, laboratories, procedures tables or discharge date from the last visit within the visit table (whichever of these activities occurs latest). This underestimated the follow-up for some patients where they were not actively using healthcare resources.

ELIGIBILITY:
Inclusion Criteria:

Included patients:

* With at least one International Classification of Diseases, 9th Revision, Clinical Modification/International Classification of Diseases,10th Revision, Clinical Modification code for PV in the identification period (01-Apr-2007 until 30-Jun-2019) that had non-missing sex and year of birth data and who were treated as part of the Integrated Delivery Network
* That were ≥ 18 years old at PV diagnosis
* With ≥ 2 prescriptions of HU
* That were classified as resistant to or intolerant of HU after a minimum of 3 months HU treatment (index date), defined as:

HCT ≥ 45% with phlebotomy (last phlebotomy within last 3 months) or Platelet count > 400 x 109/L and presence of palpable splenomegaly (palpable spleen up to 3 months after platelet count).

To identify patients in the RUX group:

- With ≥ 2 prescriptions of RUX in the post-index period.

Exclusion Criteria:

Excluded patients:

- With a MF or AML diagnosis prior to a PV diagnosis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PV patients who were resistant to or intolerant of HU in the Optum EHR database between April 2007 and June 2019
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Number of Thromboembolic events between the RUX and BAT group | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Thromboembolic events in overall Polycythemia Vera cohort and in the BAT and RUX groups were reported. A TE was defined using International Classification of Diseases 9th Revision (ICD-9- CM) and International Classification of Diseases 10th Revision (ICD-10-CM) codes previously curated as restrictive (RESPONSE RCT) and extensive (GEMFIN) definitions of TE's within the Diagnosis table in Optum EHR database.
Number of Thromboembolic events between the high and low risk subgroups of BAT group | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Within the BAT group, high risk (≥ 1 TE on average per year ) and low risk (< 1 TE on average per year) subgroups were identified based on the frequency of TEs and characterized according to patient sociodemographics, comorbidities, symptoms, clinical, and medication variables.

SECONDARY OUTCOMES:
Incidence rate of thromboembolic event | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Difference in the incidence rate of TEs in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX were reported. A TE was defined using International Classification of Diseases 9th Revision (ICD-9- CM) and International Classification of Diseases 10th Revision (ICD-10-CM) codes previously curated as restrictive (RESPONSE RCT) and extensive (GEMFIN) definitions of TE's within the Diagnosis table in Optum EHR database.
Time to first thromboembolic event | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Time to first TE in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported. A TE was defined using International Classification of Diseases 9th Revision (ICD-9- CM) and International Classification of Diseases 10th Revision (ICD-10-CM) codes previously curated as restrictive (RESPONSE RCT) and extensive (GEMFIN) definitions of TE's within the Diagnosis table in Optum EHR database.
Incidence rate of phlebotomy procedures | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Difference in the incidence rate of phlebotomies in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported.
  Phlebotomies were defined using Current Procedural Terminology, Fourth Edition (CPT4) codes within the Procedure table in Optum EHR.
Time to first phlebotomy procedure | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Time to first phlebotomy in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported. Phlebotomies were defined using Current Procedural Terminology, Fourth Edition (CPT4) codes within the Procedure table in Optum EHR.
Incidence rate of neoplasm transformations | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Difference in the incidence rate of neoplasm transformations in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported.
  A neoplasm transformation was defined as:
  * PV to MF (Myelofibrosis)
  * MF to AML (Acute Myeloid Leukemia)
  * PV to AML Neoplasm transformations were detected using ICD-9-CM and ICD-10-CM codes within the Diagnosis table in Optum EHR.
Time to first neoplasm transformation | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Time to first neoplasm transformation in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported.
  A neoplasm transformation was defined as:
  * PV to MF
  * MF to AML
  * PV to AML Neoplasm transformations were detected using ICD-9-CM and ICD-10-CM codes within the Diagnosis table in Optum EHR.
Treatment patterns: Proportion of patients using different PV-related treatments | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Differences in treatment patterns in PV patients resistant to or intolerant of HU treated with BAT compared to those treated with RUX was reported.
  BAT comprised of multiple therapies for PV including HU, IFN, pegylated IFN (PEG-IFN) and others. These therapies were reported as subcategories under BAT.
Healthcare resource utilization (HCRU): Number of inpatient hospitalizations | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Hospitalization was defined as an inpatient stay with a valid visit_ID within the Visit table in Optum EHR. Inpatient hospitalizations were reported as allcause and as PV-specific respectively
Healthcare resource utilization (HCRU): Number of outpatient visits | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Visits with the following visit type: "observation patient" with a valid visit_ID was included as an outpatient visit. Outpatient visits that resulted in an inpatient hospitalization were not included. Outpatient visits were reported as all-cause and as PV-specific respectively.
Healthcare resource utilization (HCRU): Number of emergency room visits | throughout the study, approximately 13 years (Study period: From 01-Jan-2007 to 30-Jun-2020)
  Visits with the following visit type: "emergency patient" with a valid visit_ID was included as an emergency room visit. Emergency room visits that resulted in an inpatient hospitalization were not included. Emergency room visits were reported as all-cause and as PV-specific respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CINC424B3001 from Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17945